CLINICAL TRIAL: NCT00003101
Title: A Phase II Trial of Intensive Chemotherapy and Autotransplantation for Patients With Newly Diagnosed Anaplastic Oligodendroglioma
Brief Title: Combination Chemotherapy and Bone Marrow Transplantation or Peripheral Stem Cell Transplantation in Treating Patients With Oligodendroglioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 97-077; CDR0000065833 (Registry Identifier: PDQ (Physician Data Query)); NCI-G97-1335
Record Dates: First submitted 1999-11-01; First posted 2004-05-21 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult oligodendroglioma; adult anaplastic oligodendroglioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Oligodendroglioma | interventions — Filgrastim; Busulfan; Lomustine; Procarbazine; Thiotepa; Vincristine; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: busulfan
Drug: lomustine
Drug: procarbazine hydrochloride
Drug: thiotepa
Drug: vincristine sulfate
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and combining chemotherapy with autologous bone marrow transplantation or peripheral stem cell transplantation may allow doctors to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus bone marrow transplantation or peripheral stem cell transplantation in treating patients who have oligodendroglioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the duration of response in patients with newly diagnosed pure and mixed anaplastic oligodendrogliomas treated with intensive chemotherapy supported by autologous transplantation.
* Determine the neurological and systemic toxic effects of this regimen in these patients.
* Determine the relationship of 1p loss of heterozygosity on radiographic response, progression-free survival, and overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

* Mobilization and stem cell harvest: Patients receive filgrastim (G-CSF) subcutaneously daily for up to 7 days followed by peripheral blood stem cell (PBSC) or bone marrow (BM) harvest.
* Induction therapy: All patients then receive induction therapy (PCV) comprising of oral lomustine on day 1, vincristine IV on days 8 and 29, and oral procarbazine on days 8-21. Treatment repeats every 42 days in the absence of progressive disease or unacceptable toxicity. Patients with prior complete resections receive 3 courses of PCV then proceed to high-dose chemotherapy and transplantation as described below, provided tumor has not recurred. Patients with prior partial resections or biopsies receive 2 courses of PCV and are assessed for response; those who achieve complete response (CR) or major partial response (PR) receive 1 more course of PCV. Patients who achieve partial response or have stable disease receive 2 more courses of PCV and are reassessed.
* High-dose chemotherapy and transplantation: Patients who achieve CR or PR receive thiotepa IV on days -8 to -6 and busulfan IV over 2 hours on day -5 to -3. Patients undergo autologous BM or PBSC transplantation on day 0.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study within 3-5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven anaplastic oligodendroglioma OR
* Histologically proven anaplastic mixed glioma (oligoastrocytoma) provided there is an unequivocal and substantial (at least 25%) oligodendroglial element
* No systemic or leptomeningeal metastases (excluding contiguous leptomeninges)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN) OR
* SGOT no greater than 2 times ULN

Renal

* Creatinine no greater than 1.5 times ULN

Cardiovascular

* LVEF at least 50%

Pulmonary

* DLCO at least 50% of predicted

Other

* No other serious illness that would preclude study therapy
* No other concurrent malignancy except basal cell skin cancer or carcinoma in situ of the cervix
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior systemic chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior cranial radiotherapy

Surgery

* Prior complete or partial resection, open biopsy, or stereotactic biopsy allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 1997-08; Primary Completion 2002-01 (Actual); Study Completion 2002-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M. DeAngelis, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (5):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Stanford University Medical Center, Stanford, California
  - Evanston Northwestern Health Care, Evanston, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Memorial Sloan-Kettering Cancer Center, New York, New York
- Canada (2):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario